CLINICAL TRIAL: NCT01362270
Title: Acupuncture for Sedation in the Intensive Care Unit
Brief Title: Acupuncture for Sedation in the Intensive Care Unit (ICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Jennifer M Watters, Associate Professor of Surgery, Director Surgical Critical Care, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MRF 811
Record Dates: First submitted 2011-05-25; First posted 2011-05-30 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Delirium; Respiratory Depression; Overmedication
Keywords: Anxiolytics; Sedatives; Acupuncture Therapy
MeSH Terms: conditions — Delirium; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum Acupuncture (Experimental): Subjects will receive acupuncture using real acupuncture needles.
  Interventions: Device: Verum Acupuncture
- Sham acupuncture (Sham Comparator): Subjects will receive sham acupuncture therapy using the Streitberger needle at the same points and on the same schedule as patients in the treatment group. Streitberger needles are blunt tipped and retract into themselves rather than penetrating the skin.
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Verum Acupuncture — DOSAGE: 25 acupoints per session FREQUENCY: 2 sessions per day DURATION: 5 days
  Other Names: Special No. 16 needles (Gauge 8 x 1.2")
  Arms: Verum Acupuncture
Device: Sham Acupuncture — DOSAGE: 25 acupoints per session FREQUENCY: 2 sessions per day DURATION: 5 days
  Other Names: Streitberger Placebo-needles (Gauge 8 x 1.2")
  Arms: Sham acupuncture

SUMMARY:
BACKGROUND Many patients in the trauma intensive care unit (TICU) require mechanical ventilation and sedation or anxiolysis. Mechanical ventilation means that a machine is helping a patient breathe if he can't breathe on his own. Because of the mechanical ventilation, these patients also require some medication to help keep them calm. These are called sedatives or anxiolytics.

The purpose of this study is to see if acupuncture can lower the amount of sedation and anxiolysis needed by a subject during mechanical ventilation in the TICU. Acupuncture is a medical procedure. Hair-thin sterile needles are inserted at specific points on the body.

PROCEDURES Some subjects will get acupuncture and others will get 'fake' acupuncture. By using 'fake' acupuncture, no one other than the acupuncturists will know which group a subject is in. Subjects and the team do not get to pick which subject is in which group. Instead, the groups are picked randomly. Subjects will get real or fake acupuncture twice a day for five days.

Standard of care - Both groups will receive the standard of care while in the study. They will be mechanically ventilated and given sedatives and analgesics based on the TICU protocol.

Real acupuncture group - This group will receive real acupuncture with real needles. These are stainless steel, one time use, needles. This group will also receive "ear tacks" which are like little needles that can stay on the ear for a few days. The ear tacks will be covered with a bandage so no one can tell which group the subject is in.

Sham acupuncture group - This group will receive sham needles. These needles retract into themselves much like a 'magic sword' rather than poking the skin. Subjects in this group will not get ear tacks. In order to hide the group the subject is in, a bandage will be used to cover part of the ear.

HYPOTHESIS Real acupuncture will decrease subject's sedation requirements by 30% when compared to the sham acupuncture group.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patient ≥ 18 years admitted to the Trauma ICU
* Injury Severity Score (ISS) ≥ 4
* Mechanically ventilated < 24 hours with anticipated need > 24 hours

Exclusion Criteria:

* Inability to obtain consent from patient or designee
* Receiving immunosuppressive therapy
* Receiving therapeutic anticoagulant therapy
* History of bleeding disorder, INR > 1.5, PTT > 65, PLT < 20K
* Pregnancy
* Three (3) or more inaccessible acupoints
* Head injury with elevated intracranial pressure or requiring operation
* Patients with midline abdominal incision
* Non-english speaking
* Receipt of dexmedetomidine prior to or during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Watters, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States

REFERENCES:
- [Background] Greif R, Laciny S, Mokhtarani M, Doufas AG, Bakhshandeh M, Dorfer L, Sessler DI. Transcutaneous electrical stimulation of an auricular acupuncture point decreases anesthetic requirement. Anesthesiology. 2002 Feb;96(2):306-12. doi: 10.1097/00000542-200202000-00014. PMID 11818761
- [Background] Wang SM, Kain ZN. Auricular acupuncture: a potential treatment for anxiety. Anesth Analg. 2001 Feb;92(2):548-53. doi: 10.1097/00000539-200102000-00049. PMID 11159266
- [Background] Nayak S, Wenstone R, Jones A, Nolan J, Strong A, Carson J. Surface electrostimulation of acupuncture points for sedation of critically ill patients in the intensive care unit--a pilot study. Acupunct Med. 2008 Mar;26(1):1-7. doi: 10.1136/aim.26.1.1. PMID 18356793
- [Background] McManus CA, Schnyer RN, Kong J, Nguyen LT, Hyun Nam B, Goldman R, Stason WB, Kaptchuk TJ. Sham acupuncture devices--practical advice for researchers. Acupunct Med. 2007 Jun;25(1-2):36-40. doi: 10.1136/aim.25.1-2.36. PMID 17641566
- [Background] Shapiro MB, West MA, Nathens AB, Harbrecht BG, Moore FA, Bankey PE, Freeman B, Johnson JL, McKinley BA, Minei JP, Moore EE, Maier RV; Inflammation and the Host Response to Injury Large Scale Collaborative Research Project. V. Guidelines for sedation and analgesia during mechanical ventilation general overview. J Trauma. 2007 Oct;63(4):945-50. doi: 10.1097/TA.0b013e318142d21b. No abstract available. PMID 18090028

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Verum Acupuncture | Sham Acupuncture
Started | 7 | 8
Completed | 5 | 6
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Met exclusion criteria after 1st session | 0 | 1
Not completed — Met excl. criteria before 1st session | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verum Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Success of Blinding
Description: Care team, family and subject will be surveyed to determine success of blinding. Responses will be tallied and correlated with group assignments.
Time Frame: Nurse surveyed daily for length of study (five [5] days). Physician and subject (or subject's family if he/she is unable to complete the questionnaire) surveyed upon study completion, six (6) days after enrollment.
Population: Number of participants successfully receiving assigned intervention without the care team, family, or subject knowing which treatment was given.
Measure: Count of Participants; unit: Participants
Arm/Group | Verum Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 6 | 7
Participants | 1 | 1

2. Secondary Outcome: Richmond Agitation-Sedation Scale (RAAS) Score
Description: Measure of sedation. Scale -5 to +4, with -5 equal to 'Unarousable' and +4 equal to 'Combative.'
Time Frame: Median RAAS score during treatment (5 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale from +4 to -5
Arm/Group | Verum Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 6 | 7
score on a scale from +4 to -5 | -1.4 [-3.1 to -0.4] | -1.9 [-2.8 to -0.6]

3. Secondary Outcome: Length of Ventilator Dependence
Description: Number of hours of ventilator use
Time Frame: Number hourss subject is ventilated. Subjects are expected to be ventilator dependent an average of 120 hours. Assessed up to discharge (estimated 3 weeks).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Verum Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 6 | 7
hours | 62.1 (32.4) | 232.8 (244.4)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Verum Acupuncture | Sham Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum Acupuncture (N=6) | Sham Acupuncture (N=7)
Bleeding at acupuncture site (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pain at acupuncture site (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No